CLINICAL TRIAL: NCT01582126
Title: Group Balance Training for People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro County Council (Other Government)
Collaborators: Uppsala-Örebro Regional Research Council (Other); Norrbacka-Eugenia Foundation (Other)
Responsible Party: Principal Investigator, Anette Forsberg, PhD, Researcher, RPT, Örebro County Council
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ö-1-12
Record Dates: First submitted 2012-04-16; First posted 2012-04-20 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; physical therapy; postural control
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group balance training early start (Experimental)
  Interventions: Other: Group balance training
- Group balance training late start (Experimental)
  Interventions: Other: Group balance training

INTERVENTIONS:
Other: Group balance training — Balance training i group with focus on core stability exercises and dual attention activities.

SUMMARY:
People with multiple sclerosis (MS) often have affected balance capacity and an increased risk for falls. A risk factor for falls are activities requiring dual attention. Another factor leading to reduced balance capacity is trunk stability, and decreased trunk stability has been seen in people with MS compared to healthy controls. Earlier studies using core stability exercises have shown positive effects on balance, compared to no training. In Sweden, physical therapy for people with MS has often included group training. However, evidence for this intervention is scarce. The aim of this study is therefore to investigate balance training in group. The balance training includes core stability exercises and dual attention activities. A multi-centre study is planned with a waiting-list design. Participants are randomised to either exercise group with early start or with late start. The group balance training includes training 60 minutes 2 times per week for 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed multiple sclerosis by a neurologist, being able to walk 100 m with or without walking device, being able to get down on the floor with minor assistance

Exclusion Criteria:

* No balance deficit here defined as being able to stand still heel-toe for 30 seconds with arms crossed.
* Ongoing relapse, cognitive- or language difficulties that prohibits performing the outcome measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Bergs balance scale | Change from Baseline in Bergs balance scale at 7 weeks
  Functional balance scale in sitting, standing and walking.

SECONDARY OUTCOMES:
Change from Baseline in Four Square step test | Change from Baseline in Four Square step test at 7 weeks
  Dynamic balance
Change from baseline in Timed chair stands test | Change from baseline in Times Chair stands test at 7 weeks
  Functional leg strength, rising 10 times from a chair.
Change from baseline in Timed Up and Go test | Change from baseline in Timed Up and Go test at 7 weeks
  Functional mobility.
Change from baseline in Functional Gait Assessment | Change from baseline in Functional Gait Assessment at 7 weeks
  Gait-related activities
Change from baseline in Postural sway | Change from baseline in Postural sway at 7 weeks
  Using a sway meter postural sway in standing still is assessed.
Change from baseline in Activities-specific Balance scale | Change from baseline in Activities-specific Balance scale at 7 weeks
  16 item questionnaire that includes items on balance self-efficacy
Change from baseline in 12-item Multiple Sclerosis Walking scale | Change from baseline in 12-item Multiple Sclerosis Walking scale at 7 weeks
  self-reported limitations in walking.
Change from Baseline in Bergs balance scale | Change from Baseline in Bergs balance scale at 14 weeks
  Functional balance in sitting, standing and walking
Change from Baseline in Four Square step test | Change from baseline in Four Square step test at 14 weeks
  Dynamic balance
Change from baseline in Times Chair stands test | Change from baseline in Times Chair stands test at 14 weeks
  Functional lower extremity strength
Change from baseline in Timed Up and Go test | Change from baseline in Timed Up and Go test at 14 weeks
  Functional mobility
Change from baseline in Functional Gait Assessment | Change from baseline in Functional Gait Assessment at 14 weeks
  Gait-related activities
Change from baseline in postoral sway | Change from baseline in postoral sway at 14 weeks
  Using a sway meter postural sway in standing still is assessed.
Change from baseline in Activities-specific Balance scale | Change from baseline in Activities-specific Balance scale at 14 weeks
  Balance self-efficacy
Change from baseline in 12-item Multiple Sclerosis Walking scale | Change from baseline in 12-item Multiple Sclerosis Walking scale at 14 weeks
  self-reported limitations in walking

CONTACTS AND LOCATIONS:
Overall Officials: Anette Forsberg, PhD, Study Chair — Family Medicine Research Centre, Örebro county council; Ylva Nilsagård, PhD, Principal Investigator — Centre for Health Care Sciences, Örebro county council
Locations (7):
- Sweden (7):
  - Mälarsjukhuset, Eskilstuna
  - Karlstad hospital, Karlstad
  - Rörelse och hälsa neuro, Linköping
  - Primärvård Mjölby, Mjölby
  - Nyköpings hospital, Nyköping
  - University Hospital Örebro, Örebro
  - Västerås hospital, Västerås

REFERENCES:
- [Derived] Nilsagard YE, von Koch LK, Nilsson M, Forsberg AS. Balance exercise program reduced falls in people with multiple sclerosis: a single-group, pretest-posttest trial. Arch Phys Med Rehabil. 2014 Dec;95(12):2428-34. doi: 10.1016/j.apmr.2014.06.016. Epub 2014 Jul 6. PMID 25004466